CLINICAL TRIAL: NCT05325255
Title: Effect of Myofascial Release of Subscapularis Along With Shoulder Mobilization Versus Shoulder Mobilization Alone in Adhesive Capsulitis
Brief Title: Effect of Myofascial Release of Subscapularis Along With Shoulder Mobilization in Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Umama Abbasi, Principle Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAbbasi
Record Dates: First submitted 2022-03-28; First posted 2022-04-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Adhesive capsulitis; Muscle stretching exercise; Myofascial trigger point; Range of motion; Pain
MeSH Terms: conditions — Bursitis; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland mobilization with myofascial trigger point release group (Experimental): Maitland technique: caudal, anteroposterior (AP), and posteroanterior (PA) glides 5 sets of 2-3 glides per second of Grade III and IV for 30 seconds with a rest interval of 30 second between sets.
  Ischemic Compression technique: on subscapularis trigger points for 90 secs thrice a week for 2 weeks.
  Stretching exercises in direction of abduction, external rotation (ER), internal rotation (IR), and flexion. 6 repetitions of each stretch for 10 seconds Cold pack for 20 mins
  Interventions: Other: Myofascial release of subscapularis; Other: Maitland mobilization; Other: Stretching exercises; Other: Cold pack
- Maitland mobilization alone group (Active Comparator): Maitland technique: caudal, anteroposterior (AP), and posteroanterior (PA) glides 5 sets of 2-3 glides per second of Grade III and IV for 30 seconds with a rest interval of 30 second between sets.
  Stretching exercises in direction of abduction, external rotation (ER), internal rotation (IR), and flexion. 6 repetitions of each stretch for 10 seconds Cold pack for 20 mins
  Interventions: Other: Maitland mobilization; Other: Stretching exercises; Other: Cold pack

INTERVENTIONS:
Other: Myofascial release of subscapularis — It is the application of manual pressure over myofascial trigger point that induces ischemia and causes release of trigger points
  Arms: Maitland mobilization with myofascial trigger point release group
Other: Maitland mobilization — It is the type of mobilization technique that uses passive accessory mobilization to reduce pain and stiffness and increasing range of motion
Other: Stretching exercises — It is the technique use to increase flexibility and range of motion of short and hypomobile structures
Other: Cold pack — It is the application of cold to provide analgesic effects

SUMMARY:
This randomized control trial aims to compare the effect of myofascial release of subscapularis along with shoulder mobilization VS mobilization alone among patients with adhesive capsulitis. The study will be conducted at physiotherapy outpatient department (OPD) of Sindh Institute of physical medicine and rehabilitation, and Dow University Ojha Campus, Karachi. According to study criteria, 70 patients with sub-acute adhesive capsulitis will be selected through a non-randomized purposive sampling technique by a consultant physician. After taking informed consent, participants will be randomly divided into 2 groups through the sealed envelope method. Both the groups will receive conventional treatment while Group 1 will be given an additional treatment of myofascial release of subscapularis through ischemic compression technique. Total 6 treatment sessions will be provided and assessment will be done at baseline and end of the 6th session.

DETAILED DESCRIPTION:
The sample size of 31 per group was determined using planning and specification software (PASS) version 15 software based on two independent sample t-test using 95%confidence interval and 80% power of the test. This sample was raised to 35 per group with 4 patients as drop out per group. Mean and standard deviation will be calculated for the quantitative variables while frequency and percentages will be calculated for qualitative variables. Inter-group comparison at baseline will be calculated using an independent sample t-test. The mean difference between both the techniques in terms of numeric pain rating scale (NPRS), range of motion (ROM), shoulder pain and disability index (SPADI), and pain pressure threshold(PPT) will be determined using Repeated measure 2-way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40-65 years
* Diagnosed with sub-acute adhesive capsulitis
* Pain range of 3 to 8 on NPRS
* SPADI score of >40
* Presence of myofascial trigger point in subscapularis muscle

Exclusion Criteria:

* History of fracture
* Rheumatoid arthritis
* Shoulder osteoarthritis
* Any malignancy
* Shoulder dislocation
* Subacute adhesive capsulitis with impingement syndrome

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain intensity on Numeric Pain Rating Scale in scores at 6th session (10 days) | At baseline and after 6 sessions (10 days)
  It will be use to assess pain intensity. It will be administered by simply asking the intensity of pain experienced in last 24 hours. The response of 0 represent no pain rather the responses between 1-3, 4-6, and 7-9 represents mild, moderate, and severe pain respectively. While 10 is the worst possible pain ever experienced by the person
Change from baseline joint range of motion on universal goniometer in degrees at 6th session (10 days) | At baseline and after 6 sessions (10 days)
  It will be assessed by using standard universal goniometer and measured in degrees
change from baseline shoulder disability on Shoulder pain and disability index in percentage at 6th session (10 days) | At baseline and after 6 sessions (10 days)
  Shoulder pain and disability index is used to assess shoulder disability. It consist of 13 questions i .e. 5 to assess pain and 8 to assess disability. Results will be calculated in percentage and higher results indicate increased disability. lower the percentage better will be the outcome.
Change from baseline pain pressure threshold on algometer in kilogram/centimeter2 at 6th session (10 days) | At baseline and after 6 sessions (10 days)
  assessed through algometer which provide sustained pressure from 0.05Newton/second to 20 Newton/second. Results will be recorded in kilogram/centimeter2 and higher values indicate decrease sensitivity of myofascial trigger points

CONTACTS AND LOCATIONS:
Overall Officials: Umama Abbasi, DPT, Principal Investigator — Dow University of Health Sciences; Rabail R Soomro, PhD Scholar, Study Director — Sindh Institute of Physical Medicine and Rehabilitation; Aftab Ahmed Mirza Baig, MSAPT, Study Director — Sindh Institute of Physical Medicine and Rehabilitation
Locations (2):
- Pakistan (2):
  - Sindh Institute Physical Medicine and Rehabilitation, Karachi, Sindh
  - Dow University Hospital Ojha Campus, Karachi, Sindh